CLINICAL TRIAL: NCT06266416
Title: A Family-Based HIV Prevention Program for Black Men to Protect Black Girls
Brief Title: IMARA for Black Male Caregivers and Girls Empowerment (IMAGE)
Acronym: IMAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Michigan (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Natasha Crooks, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 115207; R01MD018929 (NIH)
Record Dates: First submitted 2024-01-26; First posted 2024-02-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Sexually Transmitted Infections (Not HIV or Hepatitis); HIV Infections; Sexual Behavior
Keywords: Sexual Health; HIV Prevention; Community Based; Sexually Transmitted Infections
MeSH Terms: conditions — Sexually Transmitted Diseases; Hepatitis; HIV Infections; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: This study will evaluate the efficacy of IMAGE with 14-18-year-old Black girls (n=300) and male caregivers (n=300) in a 2-arm individually randomized controlled trial. The researchers will compare SRH outcomes (STI incidence, self-reported sexual behavior) at 6- and 12-months among girls randomized to IMAGE or a time-matched general health promotion control program (FUEL).
  The researchers will simultaneously evaluate implementation determinants (barriers, facilitators, constraints) and processes at Community Based Organizations working through the 3 steps of the implementation model (Prepare, Roll out, and Sustain).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (IMAGE) Group (Experimental): The IMAGE group will receive an 8-10-hour HIV/STI group-based (6-8 dyads) prevention program delivered to Black male caregivers and girls over 2-days.
  Interventions: Behavioral: IMARA for Black Male Caregivers and Girls Empowerment
- Control (FUEL) Group (Active Comparator): The FUEL group will receive a caregiver-adolescent general health promotion program identical in length and intensity to IMAGE.
  Interventions: Behavioral: Time-matched control program

INTERVENTIONS:
Behavioral: IMARA for Black Male Caregivers and Girls Empowerment — IMAGE is delivered by trained Black female facilitators to improve girls' SRH outcomes, prevention HIV/STIs, and reduce sexual violence. Over the two days, some components of the curriculum are delivered separately to male caregivers and girls, covering parallel content, and other sections are delivered jointly in a single group. The curriculum, extensively tailored for the target population and pilot tested, addresses Black girls' sexual development, risk for sexual violence, female anatomy, body positivity, HIV/STI knowledge and attitudes, and condom use. IMAGE is designed to strengthen bonds and communication between male caregivers and girls by encouraging perspective-taking (i.e., reverse role play) and conflict resolution.
  Other Names: IMAGE
  Arms: Experimental (IMAGE) Group
Behavioral: Time-matched control program — FUEL will engage Black male caregivers and girls to promote good nutrition, exercise, and informed consumer behavior. Topics include the impact of media on body image, evaluating nutritional labels to make healthy food choices, eating balanced meals, establishing regular exercise routines, and how families and communities can support healthy behavior. FUEL includes a brief video about HIV/AIDS and other STIs but otherwise does not otherwise address sexual health. Like IMAGE, FUEL is delivered in groups of 6-8 dyads over two workshop days (~10 hours total) in one weekend. Parts of the curriculum are delivered separately to girls and male caregivers covering parallel content and other components are delivered jointly.
  Other Names: FUEL
  Arms: Control (FUEL) Group

SUMMARY:
The scientific premise of this research is that individual, interpersonal, and structural factors impact Black girls' sexual reproductive health outcomes (sexually transmitted infection (STI) and Human Immunodeficiency Virus (HIV)) and experience of sexual violence. This study expands STI/HIV prevention programs to include Black male caregivers, a potentially valuable yet underutilized resource to protect Black girls and reduce their exposure to STI/HIV and sexual violence.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) continue to be a major public health problem for Black girls in the United States. Each year 1 in 4 Black girls, 14-19 years old acquires an STI, placing them at risk for poor sexual and reproductive health outcomes (SRH) (i.e., pelvic inflammatory disease, infertility, Human Immunodeficiency Virus (HIV)/Acquired Immunodeficiency Syndrome (AIDS)). In Chicago, STI rates are highest among 13- to 29-year-old Black girls, and they represent 56% of new HIV diagnoses compared to other racial groups, making adolescence an exceptionally vulnerable period. These racial disparities require new and innovative strategies to reduce Black girls' negative SRH outcomes. Familial protection is seen as critical to mitigating risk, particularly exposure to sexual violence, which is linked to girls' STI/HIV risk. Interventions that strengthen family relationships and communication as strategies to protect Black girls have demonstrated success in improving Black girls' SRH outcomes. Yet, with few exceptions, these programs engage only female caregivers, whereas male caregivers may amplify the protective effects of families on Black girls' SRH. The investigators systematically adapted IMARA (an evidence-based program designed for Black girls and their female caregivers) to create Informed, Motivated, Aware, and Responsible about AIDS (IMARA) for Black Male caregivers and Girls Empowerment (IMAGE), adding drivers of structural violence (i.e., stereotype messaging and lack of protection) aligning with the Becoming a Sexual Black Woman framework and the Health Disparities Research Framework. Preliminary data (interviews, focus groups, theatre, and pilot testing) with Black girls and male and female caregivers justify the proposed randomized control trial (RCT). The investigators will rigorously evaluate IMAGE's efficacy in a randomized control trial while carefully documenting implementation determinants and processes to inform adoption and sustainability. Aim 1 is to conduct a 2-arm RCT (IMAGE vs. a health promotion control) with 300 14-18-year old Black girls and their male caregivers and compare girls' sexual risk behavior (condom use, sexual debut, and sexual partners) and STI incidence at baseline, 6- and 12-months. The investigators hypothesize that girls in IMAGE will have lower STI incidence at 6- and 12- months (primary outcome) and report more condom use and fewer sexual partners (secondary outcomes) compared to the control group. The investigators will also explore change in the theoretical mechanisms posited by the Becoming a Sexual Black Woman framework. Aim 2 is to identify processes, barriers, and constraints associated with primary outcomes to inform future sustainability in community-based organizations. The long-term significance and impact of this application are high. By including Black male caregivers in the protection of girls, this study leverages a long-neglected yet important resource in Black girls' SRH, thereby amplifying the protective effects of family-based programs and pushing the science of health disparities forward.

ELIGIBILITY:
Inclusion Criteria:

AIM 1:

* Self-identify as African American, Black, or mixed race with African American or Black
* Speak English
* Males must identify as a current caregiver to girl enrolled in the study

AIM 2: All Community Based Organizations (CBO) directors and IMAGE liaisons will be eligible.

Exclusion Criteria:

AIM 1:

* Girl refuses to participate
* Inability to understand the consent/assent process
* Non-English speaking
* Does not self-identify as African American, Black, or mixed race with African American or Black
* If the primary caregiver (female caregiver/mother) does not consent to the girls' participation with the male caregiver the girl chooses, the girl will not be able to participate
* Girls will be excluded if they participated in other phases of the research

AIM 2:

• Inability to understand the consent process, and non-employment at a partnering CBO.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — AIM 1: Girls aged 14-18 years old; Male caregivers > 18 years old. AIM 2: >18 years old.
Enrollment: 612 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
STI Incidence in Participants | 6 and 12 months post treatment
  Sexually Transmitted Infection (STI) incidence from the 14-18 year old girls dyad

SECONDARY OUTCOMES:
Rate of STI History among Participants | Baseline, 6 and 12 months
  History of STI in 14-18 year old girls dyad. The investigators will ask the about a history of STI and how they have been treated.
Number of Participants Using Condoms | baseline, 6, and 12 months
  Use and frequency of condom use in 14-18 year old girls dyad
Number of Sexual Partners of Participants | baseline, 6, and 12 months
  Number of sexual partners by 14-18 year old girls dyad

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crooks N, Donenberg G, Ogwumike J, Silva J, Udeogu E, Pela E, Patil C. A randomized controlled trial of a family-based HIV/STI prevention program for Black girls and male caregivers in Chicago: IMAGE study protocol paper. PLoS One. 2025 Mar 28;20(3):e0320164. doi: 10.1371/journal.pone.0320164. eCollection 2025. PMID 40153378